CLINICAL TRIAL: NCT02970214
Title: Greifswald Approach to Individualized Medicine (GANI_MED) - Follow-up of Cardiovascular Cohorts
Brief Title: Follow-up of GANI_MED Cardio Cohorts
Acronym: GANIFU-Card
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Other Study IDs: GANIFU-C-001
Record Dates: First submitted 2016-11-09; First posted 2016-11-21 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Chronic Heart Failure; Metabolic Syndrome
Keywords: heart failure; heart disease; cardiovascular disease; metabolic risk; comorbidities
MeSH Terms: conditions — Metabolic Syndrome; Heart Failure; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — blood, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Heart Failure: Patients with chronic heart failure and with/without reduced left ventricular ejection fraction (EF) at baseline (HFrEF, HFmrEF, HFpEF)
  Interventions: Other: no intervention, only observational
- Cardiometabolic risk: Patients with cardiovascular diseases and metabolic risk factors at baseline
  Interventions: Other: no intervention, only observational

INTERVENTIONS:
Other: no intervention, only observational — no intervention, only observational

SUMMARY:
Follow-up of two hospital-based patient cohorts (heart failure, metabolic comorbidities in CVD), recruited at baseline by the GANI_MED-project (Greifswald Approach to Individualized Medicine). Standardized protocols will be used for the assessment of medical history, laboratory biomarkers, and the collection of various biosamples for bio-banking purposes. Comparisons with the general background population will be performed.

DETAILED DESCRIPTION:
5-year follow-up of two hospital-based patient cohorts (heart failure, metabolic comorbidities in CVD), recruited at baseline by the GANI_MED-project (Greifswald Approach to Individualized Medicine). Subjects will be comprehensively phenotypes using standardized protocols for the assessment of medical history, laboratory biomarkers, and the collection of various biosamples for bio-banking purposes. A multi-omics based biomarker assessment including genome-wide genotyping, transcriptome, metabolome, and proteome analyses complements the multi-level approach of GANI_MED. Comparisons with the general background population as characterized by the Study of Health in Pomerania (SHIP) will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Participation in baseline examination of GANI_MED cohorts (heart failure, metabolic risk)

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients included into the baseline examinations of the two cohorts
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2016-11; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular events | 1-year follow-ups
  Hospitalization (HF based. all-cause), myocardial infarction

SECONDARY OUTCOMES:
VO2peak | 1-year follow-ups
  Exercise capacity by CPET
QOL | 1-year follow-ups
  Quality of life by questionnaire (Minnesota Living with heart failure questionnaire)
6MW | 1-year follow-ups
  6 minute walk test distance
LVEF | 1-year follow-ups
  Left ventricular ejection fraction by echo at time of follow-up

OTHER OUTCOMES:
PWA | 1-year follow-ups
  pulse wave analysis parameters by Vascular Explorer device (neverdis GmbH, Germany)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine B, University Medicine Greifswald, Greifswald, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grabe HJ, Assel H, Bahls T, Dorr M, Endlich K, Endlich N, Erdmann P, Ewert R, Felix SB, Fiene B, Fischer T, Flessa S, Friedrich N, Gadebusch-Bondio M, Salazar MG, Hammer E, Haring R, Havemann C, Hecker M, Hoffmann W, Holtfreter B, Kacprowski T, Klein K, Kocher T, Kock H, Krafczyk J, Kuhn J, Langanke M, Lendeckel U, Lerch MM, Lieb W, Lorbeer R, Mayerle J, Meissner K, zu Schwabedissen HM, Nauck M, Ott K, Rathmann W, Rettig R, Richardt C, Salje K, Schminke U, Schulz A, Schwab M, Siegmund W, Stracke S, Suhre K, Ueffing M, Ungerer S, Volker U, Volzke H, Wallaschofski H, Werner V, Zygmunt MT, Kroemer HK. Cohort profile: Greifswald approach to individualized medicine (GANI_MED). J Transl Med. 2014 May 23;12:144. doi: 10.1186/1479-5876-12-144. PMID 24886498